CLINICAL TRIAL: NCT05069584
Title: Efficacy and Safety of Prostate Biopsies by Transperineal Versus Transrectal Route: Randomized Study
Brief Title: TransPERineal Fusion Biopsy Versus transrECTal
Acronym: PERFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A01793-38
Record Dates: First submitted 2021-09-24; First posted 2021-10-06 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transperineal biopsy (Experimental): The strategy evaluated is based on performing targeted and systematized prostate biopsies performed by the transperineal route. Biopsy must be performed as part of the usual treatment for prostate cancer diagnosis.
  Interventions: Procedure: Biopsy
- transrectal biopsy (Active Comparator): The comparison strategy is based on performing targeted and systematized prostate biopsies performed by the transrectal route. Biopsy must be performed as part of the usual treatment for prostate cancer diagnosis.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — patient must have a biopsy for his prostate cancer

SUMMARY:
Comparison of the efficacy and safety of 2 types of prostatic biopsies: transperineal biopsy versus transrectal biopsy.

DETAILED DESCRIPTION:
Interventional, comparative, randomized, controlled study in 2 parallel groups, open-label, longitudinal, multicenter, aimed at demonstrating the non-inferiority of targeted transperineal biopsies compared to targeted transrectal biopsies in terms of diagnostic efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patient having had a multiparametric prostatic MRI with the realization of 3 sequences (T2, diffusion, perfusion) interpreted by a local referent radiologist in prostate MRI or whose PI-RADS score is confirmed by rereading by a local referent radiologist in prostate MRI in case prostate MRI performed outside the center;
* Patient with at least one PI-RADS 4-5 lesion on MRI;
* Patient eligible for prostate, transperineal and transrectal biopsies, targeted and systematized;
* Patient with negative pre-biopsy antibacteriological urine examination ;
* Patient with prostate specific antigen (PSA) level ≤ 20 ng / mL;
* Patient capable of understanding the information related to the study, answering questionnaires in French, reading the instructions and having expressed their consent to participate in the study.

Exclusion Criteria:

* Patient who has already had a prostate biopsy;
* Patient with stage ≥ cT3a prostate cancer according to TNM classification version 8
* Patient with negative MRI or whose lesions have a PI-RADS score <4;
* Patient with impassable rectal stenosis;
* Patient with a dermatological disease preventing perineal access;
* Patient with rectal amputation;
* Patient presenting with a urinary tract infection;
* Patient on anticoagulant treatment at an effective oral dose, not relayed;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of the targeted biopsy in terms of detection of significant cancers. | Day 21
  Number of patients (%) diagnosed with International Society of Urological Pathology cancer grade ≥ 2 on targeted biopsies.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique La Croix Sud, Quint-Fonsegrives, France

IPD SHARING:
Plan to Share IPD: No